CLINICAL TRIAL: NCT03278691
Title: The Effect of Ketorolac on Posterior Thoracolumbar Spinal Fusions: a Prospective Randomized Controlled Trial
Brief Title: Ketorolac on Posterior Thoracolumbar Spinal Fusions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB # 1072359
Record Dates: First submitted 2017-08-24; First posted 2017-09-12 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Thoracolumbar Spinal Fusions
MeSH Terms: interventions — Sodium Chloride; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Drug: Placebo Saline 1 ml IV Q6H
  Interventions: Drug: Saline
- Intervention (Experimental): Ketorolac 15 mg (15mg/ml) IV Q6H
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Saline — 1 ml saline IV Q6H
  Arms: Placebo
Drug: Ketorolac — 15 mg (15 mg/ml) IV Q6H
  Arms: Intervention

SUMMARY:
To determine is low-dose ketorolac use in the early post-operative period (within 48 hours) provides adequate analgesia without long term adverse effect on spinal fusion rates when compared to post-operative analgesia without the use of NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Elective thoracolumbar posterior lumbar instrumented interbody fusion
* Minimally invasive spine surgery (MIS)
* 3 or fewer levels
* Bone Morphogenetic Protein (BMP) use in interbody fusion (1.05mg/level or less)
* Consent to study participation

Exclusion Criteria:

* Active tobacco smoker or history of tobacco smoking in the past 6 weeks
* Previous history of surgery at operative level(s)
* History of chronic inflammatory/rheumatological condition
* History of systemic steroid use in the past 3 months
* Auto/Workers' compensation patients
* Traumatic pathology at the operative levels
* Infection at the operative levels
* Tumor at the operative levels
* Major psychiatric illness as diagnosed by psychiatrists and on major anti- psychotic/depressants
* Patients on chemotherapeutic agents in the last 6 months
* Patients who has a history of allergy to Ketorolac
* Patients with a history of chemical addiction requiring professional rehabilitation and/or assistance
* Patients with current creatinine > 1.5mg/dl
* Patients with history of coagulopathy
* Patients with history of hepatic impairment
* Patients with uncontrolled cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fusion Construct X-Ray | 6 months postoperatively
  Each fusion level will be evaluated individually and as part of the complete fusion construct. Fusion will be evaluated by blinded independent neuroradiologists using XR.
Fusion Construct X-Ray | 12 months postoperatively
  Each fusion level will be evaluated individually and as part of the complete fusion construct. Fusion will be evaluated by blinded independent neuroradiologists using XR.
Fusion Construct X-Ray | 24 months postoperatively
  Each fusion level will be evaluated individually and as part of the complete fusion construct. Fusion will be evaluated by blinded independent neuroradiologists using XR.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) for pain | Every 8 hours x 48 hours postoperatively
  * Patient will be given the VAS on the source document in order to draw on the scale
  * Blinded investigators
Length of Stay (LOS) | 12 months postoperatively
  -Measured in days (24 hours)
  • Automatic data capture on discharge by the hospital EMR
Morphine equivalent doses | 12 months postoperatively
  -Non-study narcotics taken by patients on the floor are converted to morphine equivalent doses
  * Morphine equivalent doses are compared between the two groups daily for the first 48h
  * Data extracted from hospital EMR on discharge
Complications/Adverse events | 12 months postoperatively
  -Ketorolac-related short term in-hospital complications: GI ulceration and bleeding, GI perforation, PO bleeding, acute renal failure, anaphylactic/anaphylactoid reactions, liver failure
  * Collected by investigators daily during round
  * Document on the source document
Quality of life - long term | 12 months and/or 24 months postoperatively
  Oswestry Disability Index (ODI)
  * We will administer validated scales (ODI)
  * Face-to -face interview during clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Doris Tong, MD, Study Director — Michigan Spine and Brain Surgeons
Locations (1):
- Providence-Providence Park, Southfield, Southfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Claus CF, Lytle E, Tong D, Sigler D, Lago D, Bahoura M, Dosanjh A, Lawless M, Slavnic D, Kelkar P, Houseman C, Bono P, Richards B, Soo TM. The effect of ketorolac on posterior thoracolumbar spinal fusions: a prospective double-blinded randomised placebo-controlled trial protocol. BMJ Open. 2019 Jan 21;9(1):e025855. doi: 10.1136/bmjopen-2018-025855. PMID 30670528